CLINICAL TRIAL: NCT07241000
Title: The Efficacy of an Integrated Empowerment and Narrative Nursing Program on Enhancing Professional Identity and Alleviating Burnout Among Neonatal Nurses: A Cluster Randomized Controlled Trial
Brief Title: Integrated Program to Enhance Professional Identity and Reduce Burnout in Neonatal Nurses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Fourth Hospital of Shijiazhuang (Other)
Responsible Party: Principal Investigator, Zeyang Zhang, Principal investigator, The Fourth Hospital of Shijiazhuang
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20260974
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Professional Burnout
MeSH Terms: conditions — Burnout, Professional

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Integrated Empowerment and Narrative Nursing Program (I-ENP) Group (Experimental): Nurses in this group received a 6-month structured program in addition to usual care. The program included four monthly 2-hour empowerment education workshops and six bi-weekly 1.5-hour narrative nursing sessions, delivered in small groups.
  Interventions: Behavioral: Integrated Empowerment and Narrative Nursing Program (I-ENP)
- Control Group (Active Comparator): Nurses in this group received usual care, which included standard hospital-provided continuing education and access to employee assistance programs, without any additional specific intervention.
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Integrated Empowerment and Narrative Nursing Program (I-ENP) — A multi-component program combining empowerment education (modules on professional competence, stress management, effective communication, teamwork) and narrative nursing (sessions for story sharing, reflective writing, and peer support) delivered over 6 months.
  Arms: Integrated Empowerment and Narrative Nursing Program (I-ENP) Group
Behavioral: Usual Care — Standard hospital-provided support, including routine continuing education and access to employee assistance programs.
  Arms: Control Group

SUMMARY:
This cluster randomized controlled trial evaluates the efficacy of an integrated empowerment and narrative nursing (I-ENP) program compared to usual care for neonatal nurses. The study aims to determine if the 6-month I-ENP, which includes empowerment education and narrative nursing sessions, can enhance professional identity, reduce burnout symptoms, and lower turnover intention among neonatal nurses.

DETAILED DESCRIPTION:
Neonatal nurses are at high risk for professional burnout and weakened professional identity due to chronic workplace stressors. This study was designed to test a novel, integrated intervention combining empowerment education and narrative nursing practices. Four hospitals (clusters) were randomized to either the intervention or control group. A total of 172 neonatal nurses were included. The intervention group (n=85) participated in a structured 6-month program consisting of four empowerment education modules (covering topics like stress management and communication) and six narrative nursing sessions (involving story sharing and reflective writing). The control group (n=87) received usual care. The primary hypothesis was that the I-ENP group would show significantly greater improvement in professional identity scores compared to the control group at the end of the intervention. Secondary objectives included assessing the program's impact on burnout dimensions (emotional exhaustion, depersonalization, personal accomplishment) and turnover intention. Assessments were conducted at baseline, 6 months, and 9 months to evaluate the sustainability of the effects.

ELIGIBILITY:
Inclusion Criteria:

* Registered nurses working full-time in the Neonatal Intensive Care Units (NICUs) of the participating hospitals.
* At least 1 year of work experience.

Exclusion Criteria:

* Nurses on long-term leave (e.g., maternity leave).
* Nurses in managerial positions.
* Nurses planning to leave their position during the study period.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Change in Professional Identity Score | Baseline, 6 Months
  Change from baseline in total score on the Professional Identity Scale for Nurses (PISN). The scale ranges from 30 to 150, with higher scores indicating stronger professional identity.

SECONDARY OUTCOMES:
Change in Professional Identity Score at Follow-up | Baseline, 9 Months
  Change from baseline in total score on the Professional Identity Scale for Nurses (PISN).
Change in Burnout: Emotional Exhaustion Score | Baseline, 6 Months, 9 Months
  Change from baseline in the Emotional Exhaustion subscale score of the Maslach Burnout Inventory (MBI). Higher scores indicate greater exhaustion.
Change in Burnout: Depersonalization Score | Baseline, 6 Months, 9 Months
  Change from baseline in the Depersonalization subscale score of the MBI. Higher scores indicate greater depersonalization.
Change in Burnout: Personal Accomplishment Score | Baseline, 6 Months, 9 Months
  Change from baseline in the Personal Accomplishment subscale score of the MBI. Higher scores indicate a greater sense of personal accomplishment.
Nurse Turnover Intention | 6 Months
  Percentage of nurses reporting serious consideration of leaving their current position in the next 12 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Shijiazhuang Fourth Hospital, Shijiazhuang, Hebei, China